CLINICAL TRIAL: NCT00143221
Title: A Multicenter, Randomized, Parallel Group, Double-blind, Placebo-controlled Flexible Dose Study With and Open-label Extension to Assess the Efficacy and Safety of Viagra (Sildenafil Citrate) in the Treatment of Men With Erectile Dysfunction (ED) and Concomitant Lower Urinary Tract Symptoms (LUTS) Associated With Benign Prostatic Hyperplasia (BPH) in the United States
Brief Title: Effectiveness and Safety of Viagra in Men With ED and LUTS Due to Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481217
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Viagra
Drug: Placebo

SUMMARY:
The purpose of this study is to determine whether Viagra is effective in treating erectile dysfunction and lower urinary tract symptoms in men affected by both conditions.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of erectile dysfunction (ED)
* lower urinary tract symptoms (LUTS)

Exclusion Criteria:

* previous prostate surgery or invasive intervention for BPH
* active urinary tract disease

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2004-03; Study Completion 2005-05

PRIMARY OUTCOMES:
Comparison of change in EF domain of IIEF at Week 12 between Viagra and placebo

SECONDARY OUTCOMES:
Effect on: IPSS Effect on IPSS QoL Orgasmic Function
Sexual Desire Intercourse Satisfaction and Overall Satisfaction domains of IIEF Qmax by uroflometry
Event Log Variables

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] McVary KT, Siegel RL, Carlsson M. Sildenafil citrate improves erectile function and lower urinary tract symptoms independent of baseline body mass index or LUTS severity. Urology. 2008 Sep;72(3):575-9. doi: 10.1016/j.urology.2008.04.020. Epub 2008 Jul 2. PMID 18597830
- [Derived] McVary KT, Kaufman J, Young JM, Tseng LJ. Sildenafil citrate improves erectile function: a randomised double-blind trial with open-label extension. Int J Clin Pract. 2007 Nov;61(11):1843-9. doi: 10.1111/j.1742-1241.2007.01585.x. Epub 2007 Sep 20. PMID 17887993
- [Derived] McVary KT, Monnig W, Camps JL Jr, Young JM, Tseng LJ, van den Ende G. Sildenafil citrate improves erectile function and urinary symptoms in men with erectile dysfunction and lower urinary tract symptoms associated with benign prostatic hyperplasia: a randomized, double-blind trial. J Urol. 2007 Mar;177(3):1071-7. doi: 10.1016/j.juro.2006.10.055. PMID 17296414